CLINICAL TRIAL: NCT00822653
Title: the Effects of Plantar Stimulation on Hypotension, Treatment Efficacy and Quality of Life
Brief Title: The Effects of Plantar Stimulation on Hypotension, Treatment Efficacy and Quality of Life With Adults on Hemodialysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Original principal investigator left the university before enrollment started
Sponsor: Binghamton University (Other)
Responsible Party: Principal Investigator, Kenneth McLeod, Professor, BioEngineering, Binghamton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 521-07
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Hypotension
Keywords: hemodialysis treatment; pump stimulation; reduce hypotensive episodes
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calf Muscle Pump Stimulation (Experimental): Subjects serve as self-control. Six weeks of dialysis data without intervention will be compared to six weeks post intervention
  Interventions: Device: Calf Muscle Pump Stimulation

INTERVENTIONS:
Device: Calf Muscle Pump Stimulation — Stimulation of the postural reflex arc to activate the soleus muscle during dialysis

SUMMARY:
For the end stage renal disease (ESRD) patients undergoing hemodialysis treatment, specifically, reflex mediated calf muscle pump stimulation has the potential to significantly reduce the number and magnitude of hypotensive episodes thus enhancing the effectiveness of the dialysis process. Fewer hemodialysis complications during the patient's hemodialysis treatment, would allow treatment sessions to continue to the prescribed volume removal, with much reduced patient recovery time, and the costs associated with this recovery.

DETAILED DESCRIPTION:
Recruit individuals who consistently miss their dialysis goal. Maintain the goal over a six week period of time. Utilize exogenous calf muscle pump stimulation during each dialysis session to enhance fluid return from the lower limbs with the objective of assisting the patient in reaching ultrafiltration goal.

Track number of hypotensive events during dialysis, as well as goal success.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. alert and oriented to time, place, and self;
3. able to read and speak the English language;
4. currently receiving hemodialysis treatment approximately 3-4 hour sessions, 3 times a week;
5. received hemodialysis treatments continuously for the several previous months; AND
6. consistently exhibits hypotensive symptoms during dialysis.

Exclusion Criteria:

1. receiving hemodialysis as a temporary treatment following a peritoneal dialysis complication or an episode of transplant rejection;
2. receiving hemodialysis at home; OR
3. if they have a Medical History of any the following conditions: deep venous thrombosis, uncontrolled hypertension, pulmonary embolus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Achievement of ultrafiltration goal | 6 weeks
  Fraction of dialysis treatments where microfiltration target was achieved during 6 week period

SECONDARY OUTCOMES:
Hypotensive events | 6 weeks
  Number of hypotensive events experienced during dialysis over six week time period

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J. McLeod, Ph.D., Principal Investigator — Clinical Science and Engineering Research Center

IPD SHARING:
Plan to Share IPD: Yes
Team is willing to share anonymous data with interested investigators